CLINICAL TRIAL: NCT05619380
Title: The Effect of Manual Therapy and Therapeutic Exercises on Mandibular Analgesia, Muscles Relaxation, and Range of Motion in Patients With Masticatory Muscles Disorder
Brief Title: Effectiveness of Physiotherapy Treatments in Temporomandibular Joint Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KB-0012/102/13
Record Dates: First submitted 2022-08-24; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-08

CONDITIONS: Pain; Temporomandibular Joint Disorders; Muscle Hypertonia; Myofacial Pain; Analgesia; Musculoskeletal Pain; Craniomandibular Osteopathy
Keywords: manual therapy; physiotherapy; therapeutic exercises; masseter muscle; pain; electromyography; range of motion; temporomandibular joint
MeSH Terms: conditions — Pain; Temporomandibular Joint Disorders; Muscle Hypertonia; Facial Pain; Agnosia; Musculoskeletal Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Double (Participant,Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapeutic procedures: auto-therapy (therapeutic exercises) (Active Comparator): Specialized therapeutic exercises:
  1. Gerry's exercise - Starting position: tongue placed on the palate. Movement: slowly opening and closing the mouth. The number of repetitions: 6 times a day for 10 movements.
  2. Active lateral movements of the mandible:
     Starting position: separable teeth. Movement: slow movements of the lower jaw to the right and left. The number of repetitions: 6 times a day for 10 movements.
  3. Protrusion and mouth opening:
  Starting position: teeth separated. Movement: a) lowering the jaw forward, b) opening the mouth c) closing the mouth d) retracting the lower jaw.
  Number of repetitions: 6 times a day for 10 movements.
  Interventions: Procedure: physiotherapy treatment
- Physiotherapeutic procedures: manual therapy (massage) and auto-therapy (therapeutic exercises) (Active Comparator): Manual therapy of soft tissues in the masseter muscle:
  1. Extraoral massage of the masseter muscle (duration 5 minutes)
  2. Intraoral massage of the masseter muscle (duration 5 minutes)
  3. Functional massage of the masseter muscle (duration 5 minutes)
  Auto-therapy: The patient will receive instructions on how to perform therapeutic exercises at home.
  Interventions: Procedure: physiotherapy treatment
- Physiotherapeutic procedures: manual therapy (PIR) and auto-therapy (therapeutic exercises) (Active Comparator): Manual therapy of soft tissues in the masseter muscle:
  1. Post-isometric relaxation of the masseter muscle (duration 15 minutes).
  Auto-therapy: The patient will receive instructions on how to perform therapeutic exercises at home.
  Interventions: Procedure: physiotherapy treatment

INTERVENTIONS:
Procedure: physiotherapy treatment — Three different physiotherapy treatments will be used for, to reduce pain and tension in the masseter muscles. The assessment of pain intensity on the VAS scale will be assessed each time after the therapy. After the 5th and 10th day of therapy, it will be measured ROM and sEMG.
  Other Names: therapeutic exercises

SUMMARY:
The study will determinate the influence of four selected physiotherapeutic procedures on the pain intensity, the bioelectrical activity of the masseter muscle, and the range of mandibular mobility in patients with TMDs (temporomandibular joint dysfunction).

DETAILED DESCRIPTION:
Temporomandibular joint disorders (TMDs) are a major public health problem as they are one of the primary sources of chronic pain and impairment of chewing, swallowing, speech, and breathing function [1]. TMDs are not limited to the temporomandibular joints (TMJ) or masticatory muscles alone. Still, they are often associated with other symptoms affecting the head and neck region, such as headache, ear symptoms, and cervical spine dysfunction [1].

In recent years, there has been a significant development in the knowledge of the aetiology, diagnosis and treatment of TMDs. With the continuous search for better diagnostic and therapeutic methods, attention has begun to turn to the possibility of using non-invasive therapeutic strategies in patients with TMDs symptoms. In particular, the collaboration between dentist and physiotherapist helps in early diagnosis and improves the effectiveness of therapeutic interventions [2].

The limited number of randomised controlled trials (RCTs) comparing the efficacy of soft tissue manual therapy and self-therapy interventions prompted the researchers to focus on the analgesic and myorelaxant use of massage, post-isometric muscle relaxation (PIR) and therapeutic exercise in female patients with TMDs.

The main goals of using physiotherapy to treat TMDs are to reduce pain, reduce hypertonic muscle hyperactivity and improve tension in hypotonic muscles, restore TMJ joint mobility, and enhance mandibular proprioception and biomechanics. Physiotherapy treatment is usually reversible and non-invasive. Physiotherapy methods generally include physical techniques (laser, ultrasound, currents, heat and cold therapy), manual therapy (soft tissue therapy, joint mobilisations, massage) and therapeutic exercises. Manual therapy and therapeutic exercise in physiotherapy interventions are increasingly being used by clinicians and researched due to positive results in TMJ and some musculoskeletal problems [3].

Scientific papers show the effectiveness of masticatory muscle massage in the treatment of soft tissue disorders, achieving both muscle relaxation, improved tissue blood supply and joint range of motion and reduced pain [4]. Post-isometric relaxation (PIR) is one of the most well-known mobilisation techniques using muscle excitation and inhibition phenomena. It reduces the tension of a muscle or even an entire muscle group, as it inhibits the motoneuron field of a given muscle and thus leads to reflex relaxation. The reason for this is the activation of the Golgi tendon organs during contraction. There are 2 PIR targets - short-term and long-term. The immediate goal is primarily to combat pain and other effects of static muscle overload and to reduce muscle and connective tissue irritation. On the other hand, the long-term goal is to restore the expected length and flexibility of contracted muscles, regain normal joint range of motion and combat joint overload. As a result, post-isometric muscle relaxation is effective in, among other things, treating increased tension and reducing TrPs. It is now widely used in everyday clinical practice for both musculoskeletal therapy and TMDs.

In the daily practice of physiotherapy, it is imperative to make the patient aware of the causes and consequences of the resulting complaints and disorders. In addition to patient education, a key role is played by implementing home self-therapy into the improvement programme, mainly consisting of the systematic performance of therapeutic exercises (TE) individually selected to the patient's condition. Thanks to such management, the patient actively and consciously participates in the healing process and is taught responsibility for their own health.

ELIGIBILITY:
Inclusion Criteria:

* myofacial pain
* limited mobility of TMJ
* increased muscle tension
* Female sex

Exclusion Criteria:

* earlier splint therapy
* pharmacotherapy
* rheumatic diseases
* metabolic diseases
* fibromyalgia
* mental diseases
* pregnancy
* orthodontic treatment
* inflammation in the oral cavity
* masticatory organ injury
* lack of stability in the masticatory organ motor system

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 10 days
  Measurement on Visual Analogue Scale (VAS). It consists of a line, approximately 100 mm in length, at the left end of the scale "Score 0" witch means "no pain", at the right end of scale "Score 100mm" witch means "worst imaginable pain". The average value of all measurements will be analyzed.

SECONDARY OUTCOMES:
Electromyography surface of masseter muscle [uV- microvolts] - Rest test | 10 days
  Examination of the electrical activity of the masseter muscle at rest (Rest Test): the test will be performed on relaxed and relaxed patients. The dental arches remained slightly open during the examination. In order to eliminate the registration of signals related to the electrical activity of the eye circular muscle, these persons had their eyelids closed during the measurements. The patients were instructed not to swallow saliva during the examination and to place their tongue in a resting position. The SEMG values obtained were normalized as the ratio of RLX to MVC.
  Activity normalized to MVC [%] = Relax - RLX [µV]/ MVC [µV] x 100%
  SEMG recordings from the masseter muscles will be performed with a two-channel NeuroTrac MyoPlus 2 device with NeuroTrac software (Verity Medical Ltd., Tagoat, Ireland).
Electromyography surface of masseter muscle [uV] - maximal muscle contraction (MVC) | 10 days
  Study of the bioelectrical activity of the masseter muscle during maximal muscle contraction (MVC): SEMG signal will be recorded in a sitting position, while clenching the teeth, using the greatest possible force, within 5 seconds. The computer program with which the device cooperated registers the minimum and maximum values and calculates the average values of electric potentials. The SEMG values obtained were normalized as the ratio of RLX to MVC.
  Activity normalized to MVC [%] = RLX [µV]/ MVC [µV] x 100%
  SEMG recordings from the masseter muscles will be performed with a two-channel NeuroTrac MyoPlus 2 device with NeuroTrac software (Verity Medical Ltd., Tagoat, Ireland).

OTHER OUTCOMES:
Measurement of the range of motion (ROM) [mm] | 10 days
  Measurement of the range of mobility of the maximum abduction of the mandible (linear measurement from in mm. the upper to the lower incisor). The average value of all measurements will be analyzed.
Measurement of the range of the lateral movement of the mandible [mm] | 10 days
  Measurement of the range of mobility of the lateral movements of the mandible. The average value of all measurements will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Musculoskeletal System Rehabilitation, Pomeranian Medical University, Szczecin, Poland

REFERENCES:
- [Background] Kapos FP, Exposto FG, Oyarzo JF, Durham J. Temporomandibular disorders: a review of current concepts in aetiology, diagnosis and management. Oral Surg. 2020 Nov;13(4):321-334. doi: 10.1111/ors.12473. Epub 2020 Jan 25. PMID 34853604
- [Background] von Piekartz H, Schwiddessen J, Reineke L, Armijo-Olivio S, Bevilaqua-Grossi D, Biasotto Gonzalez DA, Carvalho G, Chaput E, Cox E, Fernandez-de-Las-Penas C, Gadotti IC, Gil Martinez A, Gross A, Hall T, Hoffmann M, Julsvoll EH, Karegeannes M, La Touche R, Mannheimer J, Pitance L, Rocabado M, Strickland M, Stelzenmuller W, Speksnijder C, van der Meer HA, Luedke K, Ballenberger N. International consensus on the most useful assessments used by physical therapists to evaluate patients with temporomandibular disorders: A Delphi study. J Oral Rehabil. 2020 Jun;47(6):685-702. doi: 10.1111/joor.12959. Epub 2020 May 4. PMID 32150764
- [Background] Daniela Biasotto-Gonzalez, Fausto Bérzin., Electromyographic study of patients with masticatory muscles disorders, physiotherapeutic treTMJent (massage), Brazilian Journal of Oral Sciences 3(10), 2004.
- [Background] Ravishankar Krishna, Anoop Sharma, Shobhit Agarwal, Sweekriti Mishra, Sanober Khan, Alternative Therapies in the Treatment of Temporomandibular Disorders, Journal of Dental & Oro-facial Research Vol. 15 , 1,2018.